CLINICAL TRIAL: NCT00944515
Title: Efficacy of Azithromycin Prophylaxis in Preventing Recurrent Acute Sinusitis in Children : A Prospective, Randomized, Double-blind, Placebo Controlled Trial.
Brief Title: Efficacy of Azithromycin Prophylaxis in Preventing Recurrent Acute Sinusitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Orathai Piboonpocanun, Department of Pediatrics, Faculty of medicine, Siriraj hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 394/2551(EC4)
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Sinusitis
Keywords: sinusitis; azithromycin
MeSH Terms: conditions — Sinusitis | interventions — Azithromycin; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azithromycin (Active Comparator): azithrimycin 3 days/week
  Interventions: Drug: azithromycin
- placebo (Placebo Comparator): placebo 3 days/week
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — placebo tablet or syrup 3 days/week
  Arms: placebo
Drug: azithromycin — azithromycin 3 days/week
  Other Names: treatment
  Arms: azithromycin

SUMMARY:
The purpose of this study is to evaluate efficacy of azithromycin prophylaxis in preventing recurrent acute sinusitis in children.

DETAILED DESCRIPTION:
A Prospective, Randomized, Double-blind, Placebo Controlled Trial of azithromycin in preventing recurrent acute sinusitis in children

ELIGIBILITY:
Inclusion Criteria:

* children between the age of 5 years and 15 years with the diagnosis of recurrent acute sinusitis who are attending the outpatient pediatric department, pediatric allergy clinic, and the ear, nose, throat clinic.

Exclusion Criteria:

* patients who have allergic rhinitis, chronic sinusitis, a history of allergic reactions to azithromycin or macrolides, treatments with immunotherapy or IVIG or gentamycin solution or pneumococcal vaccine during study period.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
frequence of acute sinusitis during 12 mouths of study period | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Orathai - Piboonpocanun, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Division of Allergy and Immunology, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No